CLINICAL TRIAL: NCT04362345
Title: Clinical Features and Risk Factors Associated With Worse Outcome in Patients Hospitalized for Covid-19 Pneumonia in France
Brief Title: Clinical Features and Risk Factors Associated With Worse Outcome in Patients Hospitalized for Covid-19 Pneumonia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7773
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-04

CONDITIONS: Covid-19
Keywords: Covid_19; SARS-CoV-2; ARDS; risk factors; infection
MeSH Terms: conditions — COVID-19; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the research is to improve patient management by rapidly identifying, based on the terrain and clinical and biological characteristics, those patients likely to present a severe form of ARDS at risk of leading to intensive care

ELIGIBILITY:
Inclusion Criteria:

* Major patient (≥18 years of age)
* Admitted in March 2020 for confirmed Covid-19 lung disease (nasopharyngeal smear or sputum with SARS-CoV-2 positive PCR).

Exclusion Criteria:

* Patient who has expressed opposition to participation in the study.
* Mild forms of infection that do not require hospitalization,
* Subject under safeguard of justice
* Subject under guardianship or trusteeship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult Patients with Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-09 (Actual); Primary Completion 2021-01-09 (Estimated); Study Completion 2021-01-09 (Estimated)

PRIMARY OUTCOMES:
Identification of risk factors for severity (death or transfer to resuscitation) of Covid-19 infection | Files analysed retrospectively from March 1st, 2020 to April 15, 2020 will be examined]

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Maladies Infectieuses et Tropicales, Strasbourg, France